CLINICAL TRIAL: NCT01529255
Title: A 3-year, Open-label, Multi-center Extension Trial of Telbivudine Therapy for Patients Previously Treated in EFFORT Clinical Trial
Brief Title: EFFORT Extension Study
Acronym: EFFORT-Ex
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Major Science and Technology Special Project of China Eleventh Five-year (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MOH-05
Record Dates: First submitted 2011-09-20; First posted 2012-02-08 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Hepatitis B, Chronic
Keywords: Chronic Hepatitis B; Compensated Chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ROADMAP (Experimental)
  Interventions: Drug: telbivudine (ROADMAP)
- SOC (Standard of Care) (Active Comparator)
  Interventions: Drug: Telbivudine (Standard of Care)

INTERVENTIONS:
Drug: telbivudine (ROADMAP) — Patients will receive oral telbivudine 600mg, daily for 104 weeks, if HBV DNA breakthrough, add on oral adefovir 10mg daily
  Stopping rules:
  The participants who achieve HBeAg seroconversion and HBV DNA<300copies/ml with over 12 months consolidation treatment in EFFORT study will discontinue treatment.
  The participants who don't meet the rules above will continue their previous treatment and follow up at the interval of 12 weeks until they finish the 156 weeks therapy or achieve the stopping rules.
  Follow up： The participants who stopped treatment will follow up at the interval of 12 weeks for 52 weeks. Of these patients, if they have confirmed virologic relapse during follow-up period, they will be excluded from the trial.
  Arms: ROADMAP
Drug: Telbivudine (Standard of Care) — Patients will receive oral telbivudine 600mg, daily for 104 weeks, if HBV DNA breakthrough, add on oral adefovir 10mg daily
  Stopping rules:
  The participants who achieve HBeAg seroconversion and HBV DNA<300copies/ml with over 12 months consolidation treatment in EFFORT study will discontinue treatment.
  The participants who don't meet the rules above will continue their previous treatment and follow up at the interval of 12 weeks until they finish the 156 weeks therapy or achieve the stopping rules.
  Follow up： The participants who stopped treatment will follow up at the interval of 12 weeks for 52 weeks. Of these patients, if they have confirmed virologic relapse during follow-up period, they will be excluded from the trial.
  Arms: SOC (Standard of Care)

SUMMARY:
* The purpose of this study is to to prove that the long-term efficacy of strategy of treatment adjustment at W24 according to virological response based on ROADMAP concept is better than standard of care strategy.
* To evaluate the off-treatment durability of HBeAg seroconversion in patients who discontinued treatment due to sustained HBeAg seroconversion and HBV DNA<300copies/ml with over 12 months consolidation treatment

ELIGIBILITY:
Inclusion Criteria:

* Treated with telbivudine or combined with adefovir in EFFORT study
* Patients are willing to participate in the extension study
* Patients provide information consent form

Exclusion Criteria:

* Adjustment of poor compliance by investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 576 (Estimated)
Dates: Start 2011-08; Primary Completion 2015-08 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The difference of percentage of patients achieving HBV DNA< 300copies/mL at week 48 in Group I and Group II | Week 48

SECONDARY OUTCOMES:
Percentage of patients achieving HBV DNA <300copies/mL at week 156 | Week 156
The log10 reduction in HBV DNA from baseline of EFFORT study at week 156 | Week 156
Percentage of patients with HBeAg loss or HBeAg seroconversion at week 156 | Week 156
Percentage of patients with HBsAg loss or HBsAg seroconversion at week 156 | Week 156
The percentage of patients with ALT normalization at week 156 | Week 156
Percentage of patients with HBV DNA breakthrough at week 156 | Week 156
Percentage of patients with genotypic resistance among the patients with HBV DNA breakthrough at week 156 | Week 156
sustained response rate of durability of HBeAg seroconversion at week 52 of off-treatment duration | week 52 of off-treatment
percentage of hepatitis flare at week 52 of off-treatment duration | week 52 of off-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jinlin Hou, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (24):
- China (24):
  - 302 Military Hospital Of China, Beijing, Beijing Municipality
  - Beijing Ditan Hospita, Beijing, Beijing Municipality
  - Beijing Friendship Hospital Attached To The Capital Medical University, Beijing, Beijing Municipality
  - BeiJing YouAn Hospital ,Capital Medical University, Beijing, Beijing Municipality
  - Department of Infectious Disease, First Hospital of Peking University, Beijing, Beijing Municipality
  - People's Hospital Under Beijnig University, Beijing, Beijing Municipality
  - The Second Affiliated of ChongQing University of Medical Science, Chongqing, Chongqing Municipality
  - Department of Infectious Disease, Nanfang Hospital, Guangzhou, Guangdong
  - No. 8 People's Hospital In GuangZhou, Guangzhou, Guangdong
  - The Third Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central-South Univrsity, Changsha, Hunan
  - No.81 Hospital of PLA, Nanjing, Jiangsu
  - First Hospital .Jilin Unniversity, Changchun, Jilin
  - ShengJing Hospital of China Medical University, Shengyang, Liaoning
  - JiNan Infectious Diseases Hospital, Jinan, Shandong
  - Changhai Hospital affiliated to Second Military Medical University, Shanghai, Shanghai Municipality
  - Huashan Hospital，Fudan University, Shanghai, Shanghai Municipality
  - No.85 Hospital of PLA, Shanghai, Shanghai Municipality
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Xian, Shanxi
  - West China Hospital.SiChuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Sixth People's Hospital of Hangzhou, Hangzhou, Zhejiang